CLINICAL TRIAL: NCT00006455
Title: International Protocol for the Treatment of Childhood Anaplastic Large Cell Lymphoma
Brief Title: Combination Chemotherapy in Treating Children With Anaplastic Large Cell Lymphoma (ALCL 99)
Acronym: ALCL 99
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Gustave Roussy, Cancer Campus, Grand Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Purpose: Treatment
Other Study IDs: CDR0000068133; FRE-IGR-ALCL99; EU-20031; NHL2000/06
Record Dates: First submitted 2000-11-06; First posted 2003-01-27 (Estimated); Last update posted 2022-05-31 (Actual); Status verified 2022-05

CONDITIONS: Lymphoma
Keywords: stage I childhood anaplastic large cell lymphoma; stage II childhood anaplastic large cell lymphoma; stage III childhood anaplastic large cell lymphoma; stage IV childhood anaplastic large cell lymphoma; recurrent childhood anaplastic large cell lymphoma
MeSH Terms: conditions — Lymphoma; Lymphoma, Large-Cell, Anaplastic | interventions — Cyclophosphamide; Cytarabine; Dexamethasone; Doxorubicin; Etoposide; Ifosfamide; Leucovorin; Methotrexate; Hydrocortisone; Vinblastine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: cyclophosphamide
Drug: cytarabine
Drug: dexamethasone
Drug: doxorubicin hydrochloride
Drug: etoposide
Drug: ifosfamide
Drug: leucovorin calcium
Drug: methotrexate
Drug: therapeutic hydrocortisone
Drug: vinblastine sulfate

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Combining more than one drug may kill more tumor cells. It is not yet known which combination chemotherapy regimen is more effective for treating anaplastic large cell lymphoma.

PURPOSE: This randomized phase III trial is studying several different regimens of combination chemotherapy to compare how well they work in treating children with anaplastic large cell lymphoma.

DETAILED DESCRIPTION:
OBJECTIVES:

* Compare the event-free survival in children with anaplastic large cell lymphoma treated with various induction and maintenance chemotherapy regimens with or without vinblastine.
* Compare the impact of different doses and schedules of methotrexate from the Berlin-Frankfurt-Munster-K2 Protocol in terms of overall survival, complete remission rate, CNS relapse rate, and nonlymphoma-related death and early death rates in these patients.

OUTLINE: This is a randomized, multicenter study. Patients are stratified according to country, vinblastine (VBL) (yes vs no), and prognostic factors (standard-risk (SR) vs high-risk (HR) disease).

Beginning immediately after confirmation of diagnosis, patients receive prephase therapy comprising dexamethasone (DM) IV or orally daily on days 1 and 2 and every 12 hours on days 3-5; cyclophosphamide (CTX) IV over 1 hour on days 1 and 2; and methotrexate (MTX) intrathecally (IT), doxorubicin (DOX) IV, and hydrocortisone (HC) IT on day 1.

Patients are then assigned to one of two treatment groups based on prognosis:

* Group 1 (SR disease): Patients are randomized to arm I or III:

  * Arm I: Patients receive treatment on arm I as defined below on day 1, and then the following courses as defined below in the following order beginning on day 6: A1, B1, A2, B2, A3, and B3.
  * Arm III: Patients receive treatment on arm III as defined below on day 1, and then the following courses as defined below in the following order beginning on day 6: regimen AM1, BM1, AM2, BM2, AM3, and BM3.
* Group 2 (HR disease):

  * First randomization: Patients are randomized to arm I or III:

    * Arm I: Patients receive treatment on arm I as defined below on day 1 and then course A1 as defined below on day 6.
    * Arm III: Patients receive treatment on arm III as defined below on day 1 and then course AM1 as defined below on day 6.
  * Second randomization: Patients without disease progression after completion of the above therapy are randomized to arm I, II, III, or IV.

    * Arm I: Patients receive treatment on arm I as defined below on day 1, and then the following courses as defined below in the following order after blood counts recover: B1, A2, B2, A3, and B3.
    * Arm II: Patients receive treatment on arm II as defined below on day 1, and then the following courses as defined below in the following order after blood counts recover: BV1, AV2, BV2, AV3, and BV3.
    * Arm III: Patients receive treatment on arm III as defined below on day 1, and then the following courses as defined below in the following order after blood counts recover: BM1, AM2, BM2, AM3, and BM3.
    * Arm IV: Patients receive treatment on arm IV as defined below on day 1, and then the following courses as defined below in the following order after blood counts recover: BMV1, AMV2, BMV2, AMV3, and BMV3.

Patients are followed every 2 months for 1 year, every 4 months for 2 years, every 6 months for 2 years, and then annually thereafter.

DEFINITIONS:

* Arms I-IV are defined below:

  * Arm I: Patients receive lower dose MTX IV over 24 hours and MTX IT.
  * Arm II: Patients receive lower dose MTX IV over 24 hours and MTX IT. Patients with HR disease also receive VBL IV weekly for 1 year beginning 3 weeks after initiation of course BV3.
  * Arm III: Patients receive higher dose MTX IV over 3 hours without intrathecal therapy.
  * Arm IV: Patients receive treatment as in arm III. Patients with HR disease also receive VBL IV weekly for 1 year beginning 3 weeks after initiation of course BMV3.
* Regimens A, B, AV, BV, AM, BM, AMV, and BMV are defined below:

  * Regimen A (courses A1, A2, and A3): Patients receive DM IV or orally every 12 hours on days 1-5; MTX IV over 24 hours on day 1; MTX IT, DOX IV and HC IT (beginning 2-4 hours after initiation of MTX infusion) on day 1; leucovorin calcium (CF) IV rescue at 42, 48, and 54 hours after initiation of MTX infusion; ifosfamide (IFF) IV over 1 hour on days 1-5 (before initiation of MTX infusion); cytarabine (ARA-C) IV over 1 hour every 12 hours and etoposide (VP-16) IV over 2 hours once (beginning after completion of ARA-C infusion) on days 4 and 5. Each course lasts 3 weeks.
  * Regimen B (courses B1, B2, and B3): Patients receive DM, MTX, intrathecal therapy, and CF rescue as in regimen A. Patients also receive CTX IV over 1 hour on days 1-5 and DOX IV over 1 hour on days 4 and 5. Each course lasts 3 weeks.
  * Regimen AV (courses AV1, AV2, and AV3): Patients receive treatment as in regimen A and VBL IV on day 1. Each course lasts 3 weeks.
  * Regimen BV (courses BV1, BV2, and BV3): Patients receive treatment as in regimen B and VBL IV as in regimen AV. Each course lasts 3 weeks.
  * Regimen AM (courses AM1, AM2, and AM3): Patients receive DM IV or orally every 12 hours on days 1-5; MTX IV over 3 hours on day 1; and CF IV rescue every 6 hours for a total of 12 doses beginning 24 hours after initiation of MTX infusion. Patients also receive IFF, ARA-C, and VP-16 as in regimen A. Each course lasts 3 weeks.
  * Regimen BM (courses BM1, BM2, and BM3): Patients receive CTX and DOX as in regimen B. Patients also receive DM, MTX, and CF rescue as in regimen AM. Each course lasts 3 weeks.
  * Regimen AMV (courses AMV1, AMV2, and AMV3): Patients receive treatment as in regimen AM and VBL as in regimen AV. Each course lasts 3 weeks.
  * Regimen BMV (courses BMV1, BMV2, and BMV3): Patients receive treatment as in regimen BM and VBL as in regimen AV. Each course lasts 3 weeks.

PROJECTED ACCRUAL: A total of 400 patients will be accrued for this study within 5.4-6.7 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically proven standard-risk (SR) or high-risk (HR) anaplastic large cell lymphoma

  * SR disease defined by no involvement of the skin, mediastinum, liver, spleen, or lung
  * HR disease defined by any of the following:

    * Biopsy proven skin lesions (except skin lesions overlying an involved node or isolated skin disease)
    * Mediastinal involvement by x-ray or CT scan
    * Involvement of the liver (enlarged by at least 5 cm and/or nodular), spleen (enlarged and/or nodular), or lung (biopsy not needed for obvious lesions)
* Histologic or cytologic slides must be available for national pathology review for all patients not meeting the classical criteria for diagnosis (typical histopathology, immunohistochemistry: CD30 positive, endomysial antibody positive, nucleophosmin negative, anaplastic lymphoma kinase (ALK) positive (if available), null or T-immunophenotype) unless proven t(2;5)
* Must enroll within 1 week prior to beginning study regimen A
* No CNS involvement (CSF or cerebral tumor)
* First randomization (SR or HR disease):

  * Must have begun prephase therapy
  * No isolated primary skin disease
  * No low-risk disease defined as completely resected stage I disease
* Second randomization (HR disease only):

  * Must have completed first randomization therapy without disease progression

PATIENT CHARACTERISTICS:

Age:

* Under 22

Performance status:

* Not specified

Life expectancy:

* Not specified

Hematopoietic:

* See Disease Characteristics

Hepatic:

* See Disease Characteristics

Renal:

* Not specified

Pulmonary:

* See Disease Characteristics

Immunologic:

* No congenital immunodeficiency
* No AIDS

Other:

* No prior malignancy

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* Not specified

Chemotherapy:

* Not specified

Endocrine therapy:

* Prior corticosteroids for anaplastic large cell lymphoma allowed if given for no more than 8 days

Radiotherapy:

* Not specified

Surgery:

* No prior organ transplantation

Other:

* No other prior therapy for anaplastic large cell lymphoma

Ages: 0 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 885 (Actual)
Dates: Start 1999-11-26 (Actual); Primary Completion 2009-01-12 (Actual); Study Completion 2020-09-03 (Actual)

PRIMARY OUTCOMES:
Event-free survival

SECONDARY OUTCOMES:
Overall survival
Complete remission achieved after treatment course B3 and lasting ≥ 4 weeks
Short- and long-term toxicity
Nonlymphoma related death and early deaths (excluding deaths occurring after second-line treatment for failure or relapse)
CNS relapses

CONTACTS AND LOCATIONS:
Overall Officials: Laurence Brugieres, MD, Study Chair — Gustave Roussy, Cancer Campus, Grand Paris
Locations (10):
- St. Anna Children's Hospital, Vienna, Austria
- U.Z. Gasthuisberg, Leuven, Belgium
- Institut Gustave Roussy, Villejuif, France
- Kinderklinik, Giessen, Germany
- Azienda Ospedaliera di Padova, Padua, Italy
- Dutch Childhood Leukemia Study Group, The Hague, Netherlands
- Hospital Clinico Universitario de Valencia, Valencia, Spain
- Karolinska University Hospital - Huddinge, Stockholm, Sweden
- University Children's Hospital, Zurich, Switzerland
- Addenbrooke's Hospital, Cambridge, England, United Kingdom

REFERENCES:
- [Result] Attarbaschi A, Mann G, Rosolen A, Williams D, Uyttebroeck A, Marky I, Lamant L, Horibe K, Wrobel G, Beishuizen A, Wossmann W, Reiter A, Mauguen A, Le Deley MC, Brugieres L; European Intergroup for Childhood Non-Hodgkin Lymphoma (EICNHL) ALCL99 Trial. Limited stage I disease is not necessarily indicative of an excellent prognosis in childhood anaplastic large cell lymphoma. Blood. 2011 May 26;117(21):5616-9. doi: 10.1182/blood-2010-12-324012. Epub 2011 Mar 28. PMID 21444917
- [Result] Wrobel G, Mauguen A, Rosolen A, Reiter A, Williams D, Horibe K, Brugieres L, Le Deley MC; European Inter-Group for Childhood, Non-Hodgkin Lymphoma (EICNHL). Safety assessment of intensive induction therapy in childhood anaplastic large cell lymphoma: report of the ALCL99 randomised trial. Pediatr Blood Cancer. 2011 Jul 1;56(7):1071-7. doi: 10.1002/pbc.22940. Epub 2011 Jan 28. PMID 21280197
- [Result] Le Deley MC, Rosolen A, Williams DM, Horibe K, Wrobel G, Attarbaschi A, Zsiros J, Uyttebroeck A, Marky IM, Lamant L, Woessmann W, Pillon M, Hobson R, Mauguen A, Reiter A, Brugieres L. Vinblastine in children and adolescents with high-risk anaplastic large-cell lymphoma: results of the randomized ALCL99-vinblastine trial. J Clin Oncol. 2010 Sep 1;28(25):3987-93. doi: 10.1200/JCO.2010.28.5999. Epub 2010 Aug 2. PMID 20679620